CLINICAL TRIAL: NCT04921085
Title: Nutritional Status Study of Inpatients in Hospitals
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang University (Other); Zhejiang Provincial People's Hospital (Other); The Second Affiliated and Yuying Children's Hospital of Wenzhou Medical University (Unknown); Sir Run Run Shaw Hospital (Other); Red Cross Hospital, Hangzhou, China (Other); Jinhua Municipal Central Hospital (Other); Quzhou People' s Hospital (Unknown); The Central Hospital of Lishui City (Other); Lishui People' s Hospital (Unknown); Jinhua People' s Hospital (Unknown); Yuyao People's Hospital (Other); Ningbo No. 1 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Zhejiang Hospital (Other); Huizhou Municipal Central Hospital (Other); The First People's Hospital of Huzhou (Other); Cancer Hospital of The University of Chinese Academy of Sciences (Unknown); Hangzhou Medical College (Other); Zhejiang Provincial Tongde Hospital (Other); Shaoxing People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-928
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-04

CONDITIONS: Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult inpatients: adult inpatients with 7 categories of diseases (including digestive system, respiratory system, cardiovascular and endocrine system, tumor, nervous system, and urinary system)
  Interventions: Other: Cross-sectional obeservational survey

INTERVENTIONS:
Other: Cross-sectional obeservational survey — Cross-sectional obeservational survey

SUMMARY:
evaluating the nutritional status of inpatients with 7 catogories of diseases ( including digestive system, respiratory system, cardiovascular and endocrine system, tumor, nervous system, urinary system) within 24~48 hours after admission. Among them, the Second Affiliated Hospital of Zhejiang University School of Medicine has undertaken 200 cases, and a total of 25 hospitals in zhejiang participated（5000 cases in total）.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with 7 categories of diseases (including digestive system, respiratory system, cardiovascular and endocrine system, tumor, nervous system, and urinary system)
* Age ≥ 18
* 24～48h after admission

Exclusion Criteria:

* Age<18
* Critically ill patient
* With mental illness and cannot think or behavior normally
* Any other serious or uncontrolled illness which the investigator think is undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult inpatients with within 7 categories of diseases (including digestive system, respiratory system, cardiovascular and endocrine system, tumor, nervous system, and urinary system)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Nutritional risk screening scored with NRS 2002 questionnaire | 24~48 hours after admission
  Detect the presence of undernutrition and the risk of developing undernutrition by Risk Screening 2002 questionnaire(NRS-2002) . The overall score range is from 0 to 7, when score≥3, the patient is nutritionally at-risk

SECONDARY OUTCOMES:
Body fat mass | 24~48 hours after admission
  Body Fat Mass is assessed by bioelectrical impedance analysis (BIA)
Body muscle mass | 24~48 hours after admission
  Body muscle mass is assessed by bioelectrical impedance analysis (BIA)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China